CLINICAL TRIAL: NCT00630240
Title: Investigation the Risk Factors for the Leakage of Anticancer Drugs to Systemic Circulation in Patients With Hepatocellular Carcinoma Treated by Transcatheter Arterial Chemoembolization
Brief Title: Risk Factors for the Leakage of Anticancer Drugs to Systemic Circulation by Transcatheter Arterial Chemoembolization
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Zu-Yau Lin/ Kaoshing Medical University Chung-Ho Memorial Hospital, Kaoshing Medical University Chung-Ho Memorial Hospital
Other Study IDs: KMUH-IRB-960297; KMUH-IRB-960297
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: epirubicin; mitomycin C; cisplatin; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: only one arm for study

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common malignant tumor of the liver. Transcatheter arterial chemoembolization (TACE) is the traditional method for the palliative management of patients with HCC. Few previous studies had demonstrated that the serum level of anticancer drug from patients treated by TACE was similar to those treated by systemic chemotherapy. The defense ability of the patient treated by TACE may thus be influenced by the leakage of anticancer drug to the systemic circulation. Since more than 80% patients with HCC also have liver cirrhosis, the toxicity for those anticancer drugs with hepatic transformation will be increased caused by the cirrhotic liver. The severity of pancytopenia in cirrhosis will be exacerbated by the effect of bone marrow suppression caused by anticancer drugs. Patients are at high risk for infection and hemorrhage. Therefore, it is of clinical importance to prevent or decrease the leakage of anticancer drugs to systemic circulation in patients treated by TACE. The procedures of TACE performed by previous studies were not constant and the distributions of tumor vessels were not evaluated in detail. The possible risk factors for the leakage of anticancer drug have not been investigated. This project will collect 60 patients with HCC including 30 patients with hepatitis B and 30 patients with hepatitis C. The blood levels of anticancer drugs (epirubicin, mitomycin C and cisplatin) will be determined within one hour and at the third day after TACE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatocellular carcinoma caused by hepatitis B or C who will be treated by TACE

Exclusion Criteria:

* Previously treated by antiviral drugs for hepatitis B or C

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hepatocellular carcinoma caused by hepatitis B or C
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The blood levels of anticancer drugs (epirubicin, mitomycin C and cisplatin) will be determined within one hour and at the third day after TACE. | within one hour and at the third day after TACE

CONTACTS AND LOCATIONS:
Overall Officials: z y lin, MD, Ms, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Division of Hepatobiliary Medicine, Department of Internal Medicine, Kaohsiung Medical University Hospital, No. 100 Tzyou 1st Road, Kaohsiung City, Taiwan